CLINICAL TRIAL: NCT01032811
Title: Pilot Study Of Primary And Secondary Attention-Deficit/Hyperactivity Disorder Among Survivors Of Childhood Cancer
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SADHD1
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: ADHD; Cancer
Keywords: ADHD, childhood cancer; ADHD/Secondary ADHD Among Survivors of Childhood Cancer
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Participants: St. Jude Children's Research Hospital patients from Leukemia, Neuro-Oncology, Radiation Oncology, and After Completion of Therapy (ACT) clinics.

SUMMARY:
This is a pilot study that will be an exploratory investigation of the rate of occurrence of ADHD/S-ADHD in adolescent cancer survivors. The procedures that will be used for identifying attention problem symptoms, determining the frequency and severity of such symptoms, and characterizing the level of impairment resulting from the symptoms are novel to pediatric oncology research.This pilot study will draw from the approach used in traumatic brain injury research of post-injury effects to illuminate more clearly the nature of attentional late effects experienced by survivors of childhood cancer.

DETAILED DESCRIPTION:
1. This study will investigate the feasibility of assessing symptoms of developmental ADHD and "secondary ADHD" (S-ADHD) among adolescent survivors of childhood cancer using a structured diagnostic clinical interview procedure. (S-ADHD describes an acquired clinical presentation that is consistent with the diagnostic criteria of ADHD).
2. This study will provide preliminary estimates of the rate of occurrence of ADHD/S-ADHD among adolescent survivors of childhood cancer as compared to the prevalence of developmental ADHD in the general population.
3. The study will examine the relationship between ADHD/S-ADHD symptoms and laboratory measures traditionally used to assess specific components of attention (e.g., CPT) in survivors of childhood cancer.
4. The study will examine the relationship between ADHD/S-ADHD symptoms and smoking (including intentions, behaviors, and motivators) among adolescent survivors of childhood cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated for acute lymphoblastic leukemia (ALL) OR primary central nervous system (CNS) tumor.
2. Completed primary treatment at least one year prior to enrollment with no evidence of active disease.
3. Age 12-17 years inclusive at the time of enrollment.
4. At least one parent/guardian must be present.
5. Participant and parent are able to understand English.
6. Participant and parent are willing and able to provide consent/assent according to institutional guidelines.
7. Parent/guardian signs consent.

Exclusion Criteria:

1.Significant impairment in intellectual functioning (e.g., full or estimated IQ <70) as documented in the medical record.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited through consecutive enrollment in the SJCRH Leukemia, Neuro-Oncology, Radiation Oncology, and After Completion of Therapy (ACT) clinics. Participants will be accrued using a broad stratification process for gender (female, male) and age (12-14 years, 15-17 years) for each diagnosis group (brain tumor, ALL).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
This study will investigate the feasibility of assessing symptoms of developmental ADHD and "secondary ADHD" (S-ADHD) among adolescent survivors of childhood cancer using a structured diagnostic clinical interview procedure. | 1 year
This study will provide preliminary estimates of the rate of occurrence of ADHD/S-ADHD among adolescent survivors of childhood cancer as compared to the prevalence of developmental ADHD in the general population. | 1 year

SECONDARY OUTCOMES:
This study will examine the relationship between ADHD/S-ADHD symptoms and laboratory measures traditionally used to assess specific components of attention (e.g., CPT) in survivors of childhood cancer. | 1 year
This study will examine the relationship between ADHD/S-ADHD symptoms and smoking (including intentions, behaviors, and motivators) among adolescent survivors of childhood cancer. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sean Phipps, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: Related Info — http://www.stjude.org